CLINICAL TRIAL: NCT02868008
Title: The Efficacy of Multimodal Magnetic Resonance Imaging Techniques in Assessing the Surgical Risk for Eloquent Arteriovenous Malformations
Brief Title: Multimodal Imaging Techniques in Assessing the Surgical Risk for Eloquent Arteriovenous Malformations
Acronym: MITASREAVM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Chinese PLA General Hospital (Other); Beijing Hospital (Other Government); Xuanwu Hospital, Beijing (Other); Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Dr. Yong Cao, Professor, Beijing Tiantan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCW2016-11-AVM
Record Dates: First submitted 2016-07-25; First posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Intracranial Arteriovenous Malformations
Keywords: multimodal imaging; surgical risk; arteriovenous malformations
MeSH Terms: conditions — Intracranial Arteriovenous Malformations; Arteriovenous Malformations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- fMRI guided AVM resection (Experimental): fMRI guided microsurgical resection of brain AVMs
  Interventions: Procedure: Microsurgical resection of brain AVMs

INTERVENTIONS:
Procedure: Microsurgical resection of brain AVMs — fMRI guided microsurgical resection of brain AVMs

SUMMARY:
Microsurgical resection for eloquent arteriovenous malformations (AVMs) remains challenging. Currently, there are only two grading systems concerning pretreatment assessment of brain AVMs: the Spetzler-Martin grading system proposed by Spetzler and Martin in 1986 and the supplementary grading system proposed by Lawton in 2010. Controversies exist regarding the treatment timing and treatment modalities for eloquent AVMs. Till now, there is no clinical trial concerning the efficacy of multimodal magnetic resonance imaging techniques in assessing the surgical risk for eloquent AVMs. The investigators assume that multimodal imaging-based grading system is superior to the classic Spetzler-Martin grading system and the supplementary grading system in predicting the surgical risk for eloquent AVMs.

DETAILED DESCRIPTION:
Microsurgical resection for eloquent arteriovenous malformations (AVMs) remains challenging. Currently, there are only two grading systems concerning pretreatment assessment of brain AVMs: the Spetzler-Martin grading system proposed by Spetzler and Martin in 1986 and the supplementary grading system proposed by Lawton in 2010. Controversies exist regarding the treatment timing and treatment modalities for eloquent AVMs. Till now, there is no clinical trial concerning the efficacy of multimodal magnetic resonance imaging techniques in assessing the surgical risk for eloquent AVMs. The investigators assume that multimodal imaging-based grading system is superior to the classic Spetzler-Martin grading system and the supplementary grading system in predicting the surgical risk for eloquent AVMs.

This study consists of two parts: a retrospective analysis and a prospective study. Firstly, the investigators will retrospectively review the 250 AVM patients that were surgically treated at Beijing Tiantan Hospital between June 2012 and June 2015. All data of these patients were prospectively maintained in our AVM database. All these patients had preoperative functional magnetic resonance imaging (fMRI) studies. The investigators will collect the patient demographic data, AVM features, the least distances from the AVMs to the activated cortex as well as to the fiber tracts. The investigators will also collect the patient preoperative functional status (modified Rankin scale score, mRS) and the functional status (mRS) six months after surgery. The changes between the two functional status in mRS will be classified into two groups: those with worsened mRS (mRS score six months after surgery - presurgical mRS score >0) and those with unchanged or improved mRS (mRS score six months after surgery - presurgical mRS score ≤0). The new grading system will be proposed based on the multimodal magnetic resonance imaging (MRI). The investigators will compare the predictive accuracy of the three grading systems (the Spetzler-Martin grading system, the supplementary system and our new grading system) in assessing functional status (worsened mRS). Then in the prospective study, the investigators will enroll 400 surgically treated AVM patients from five neurosurgical centers. All patients will meet the inclusion and exclusion criteria. The preoperative preparation, the surgical procedures, the follow-up period, the primary outcomes and statistical analyses will be the same as those in the retrospective study part. Multimodal imaging-based system will be verified in this prospective phase. If the results demonstrate that the multimodal MRI-based grading system is superior to the Spetzler-Martin grading system and the supplementary system in predicting the functional status six months after AVM surgery, the investigators will propose the new AVM grading system in the public.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 12 and 60 years
2. Data from preoperative structural MRI, blood oxygen level dependent (BOLD)-fMRI, time-of-flight magnetic resonance angiography (TOF-MRA), and DTI of the motor tract,language tract or optic radiation were available
3. Patients with a definite diagnosis of AVM confirmed by preoperative digital subtraction angiography
4. Patients opting for surgical management at the five centers in this study
5. Patients without any interventional therapy (microsurgery, radiosurgery, endovascular embolization, or multimodality treatment) before admission to the five centers

Exclusion Criteria:

1. Patients with acute intracranial hematoma and resultant brain hernia prompting emergency surgery
2. Patients with a hemorrhagic incident in the past month
3. Nonavailability of BOLD-fMRI and DTI data
4. Patients with other severe diseases that prevented them from having surgery
5. Patients unwilling to participate in the trial

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
neurologic status measured by modified Rankin scale score | six months after AVM surgery
  the changes of modified Rankin scale (mRS) score six months after AVM surgery compared with the presurgical mRS score

SECONDARY OUTCOMES:
number of patient deaths | within 6 months after surgery
  number of patient deaths due to AVM rebleeding or surgery
AVM obliteration confirmed by postoperative DSA or CTA | within one week after surgery
  AVM obliteration on DSA or CTA
AVM rebleeding confirmed by CT scan | within 6 months after surgery
  AVM rebleeding confirmed by CT scan within 6 months after surgery
Seizure control measured by Engel classification | within 6 months after surgery
  Seizure control or new seizure onset according to Engel classification within 6 months after surgery
muscle strength measured by muscle strength grading scale | 6 months after surgery
  muscle strength according to muscle strength grading scale 6 months after surgery
number of patients with aphasia | 6 months after surgery
  number of patients with aphasia measured by Western Aphasia Battery (WAB) 6 months after surgery
number of patients with visual field defect | 6 months after surgery
  number of patients with visual field defect measured by visual field testing 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Shuo Wang, M.D., Study Chair — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wen Z, Zheng K, Guo S, Liu Y, Wang K, Liu Q, Wu J, Wang S. The difference of functional MR imaging in evaluating outcome of patients with diffuse and compact brain arteriovenous malformation. Neurosurg Rev. 2024 Jul 24;47(1):347. doi: 10.1007/s10143-024-02593-9. PMID 39043982
- [Derived] Jiao Y, Lin F, Wu J, Li H, Fu W, Huo R, Cao Y, Wang S, Zhao J. Plasticity in language cortex and white matter tracts after resection of dominant inferior parietal lobule arteriovenous malformations: a combined fMRI and DTI study. J Neurosurg. 2020 Mar 20;134(3):953-960. doi: 10.3171/2019.12.JNS191987. Print 2021 Mar 1. PMID 32197246
- [Derived] Li M, Jiang P, Guo R, Liu Q, Yang S, Wu J, Cao Y, Wang S. A Tractography-Based Grading Scale of Brain Arteriovenous Malformations Close to the Corticospinal Tract to Predict Motor Outcome After Surgery. Front Neurol. 2019 Jul 17;10:761. doi: 10.3389/fneur.2019.00761. eCollection 2019. PMID 31379715
- [Derived] Tong X, Wu J, Cao Y, Zhao Y, Wang S. New predictive model for microsurgical outcome of intracranial arteriovenous malformations: study protocol. BMJ Open. 2017 Jan 27;7(1):e014063. doi: 10.1136/bmjopen-2016-014063. PMID 28132013